CLINICAL TRIAL: NCT06812923
Title: The Study on Effectiveness and Mechanisms of Transcranial Alternating Current Stimulation in Treating Increased Inflammatory Activity Refractory Depression
Brief Title: TACS on High-inflammatory and Refractory Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Principal Investigator, Jie Li, professor, Tianjin Anding Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJAD-tACS15
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Treatment Resistant Depression (TRD); Inflammation
Keywords: treatment resistant depression; transcranial Alternating Current Stimulation; C-reactive protein
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Inflammation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tACS group (Experimental): participants receive tACS (15mA、77.5Hz tACS) treatment for 20 times (5 times a week, four weeks totally), with ongoing antidepressant treatment.
  Interventions: Device: transcranial Alternating Current Stimulation (tACS)
- Sham group (Sham Comparator): participants receive sham stimulation for 20 times (5 times a week, four weeks totally), with ongoing antidepressant treatment.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: transcranial Alternating Current Stimulation (tACS) — tACS, parameters: 15mA、77.5Hz tACS, 20 times (5 times a week, four weeks totally)
  Arms: tACS group
Device: Sham stimulation — Sham stimulation, matched with real tACS, except for providing electrical stimulation
  Arms: Sham group

SUMMARY:
This study is a randomized controlled trial with a duration of 12 weeks (4 weeks of intervention + 8 weeks of follow-up). The participants are patients with treatment-resistant depression (TRD) and high inflammatory activity (n=52). The study aims to clarify the effectiveness of 15mA, 77.5Hz transcranial alternating current stimulation (tACS) in treating TRD with high inflammatory activity by comparing the changes in depressive symptoms and biological markers after active tACS stimulation versus sham stimulation. Additionally, the study seeks to explore potential underlying mechanisms of action.

DETAILED DESCRIPTION:
This experiment is a randomized controlled trial lasting 12 weeks (4 weeks of intervention + 8 weeks of follow-up), with participants being patients with treatment-resistant depression (TRD) and high inflammatory activity (n=52). The study aThis study plans to include 52 patients with treatment-resistant depression (TRD) and high inflammatory activity who meet the inclusion and exclusion criteria. Participants will be randomly assigned to either the active stimulation group (active group, n=26) or the sham stimulation group (sham group, n=26). During the baseline phase, basic information (e.g., gender, age, age of onset, family history of mental illness) will be collected, and assessments using scales (as detailed in the experimental methods) will be completed. EDTA blood collection tubes will be used to collect 10ml of fasting peripheral venous blood (-80°C for storage). The intervention will begin the following day with either tACS or sham stimulation.

Before the first tACS or sham treatment, participants will undergo resting-state electroencephalogram (EEG) recordings to assess brain wave activity in different brain regions. Participants will receive a total of 20 sessions of tACS or sham intervention (5 sessions per week, with a break on weekends). At the end of weeks 2 and 4, the scales will be reassessed. After the 4-week intervention period ends, another EEG will be recorded, and fasting peripheral venous blood (10ml) will be collected the following morning for storage.

After the intervention phase, participants will enter an 8-week follow-up period. At the 8th and 12th weeks, all participants will undergo a reassessment using the HAMD-17 scale and provide 10ml of peripheral venous blood for analysis. The data from the scales, blood analysis, and EEG will be summarized and used for statistical analysis. Throughout the study, participants' antidepressant medication will remain unchanged.

The specific details are as follows:

1. Assessment of Treatment Efficacy:

   The changes in depressive symptoms before and after treatment will be compared within groups using the HAMD-17 scale, allowing the quantification of the clinical effect of tACS treatment. Between-group comparisons will be made between the active tACS group and the sham stimulation group to evaluate the difference in actual therapeutic efficacy versus placebo effect.
2. Analysis of Changes in Peripheral Blood Biomarkers:

   Blood samples will be analyzed for levels of inflammatory factors and glial cell activity markers before and after treatment. This will help explore the correlation between these biomarkers and depressive symptoms. It may provide insights into whether the antidepressant effects of tACS are mediated by biological changes, specifically whether tACS works by modulating immune-inflammatory responses.
3. Assessment of Electroencephalogram (EEG) Changes:

   EEG recordings will be analyzed to assess brain wave activity in different brain regions before and after treatment. This will help explore the relationship between changes in brain wave power in specific regions and the improvement in depressive symptoms, as well as how these changes relate to the levels of biological markers.
4. Long-Term Follow-Up Results:

   Follow-up at 8 weeks and 12 weeks after treatment will provide data on the durability of the tACS treatment effect. This will help assess the potential long-term value of tACS in the management of treatment-resistant depression.
5. Insights into Mechanisms of Action and Etiology:

The models established through data analysis may reveal how tACS affects the underlying etiology of depression, particularly the role of immune-inflammatory responses. These insights could help identify new therapeutic targets for treatment-resistant depression and facilitate the development of novel treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged between 18 and 55 years; (2) Diagnosed with depression through a structured clinical interview by a psychiatrist using the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); (3) A total score of 17 or above on the 17-item Hamilton Depression Rating Scale (HAMD-17), with a score of 2 or more on item 1 (depression); (4) CRP level between 0.85-10 mg/L; (5) DM-TRD score of at least 12.5; (6) Stable use of treatment medications (antidepressants, antipsychotics) for at least 2 weeks during the current depressive episode; (7) Able to understand and sign the informed consent form.

Exclusion Criteria:

* (1) A history of current or past seizures, epilepsy, hydrocephalus, central nervous system tumors, or acute brain injury and infections; (2) A score of 3 or 4 on item 3 of the HAMD-17, or a history of suicidal behavior with significant suicide risk; (3) Received electroconvulsive therapy (ECT), modified electroconvulsive therapy (MECT), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), tACS, or other neuromodulation treatments within one month prior to enrollment; (4) Pregnant or breastfeeding women; (5) Patients with any severe organic disease or in an unstable condition due to organic disease; (6) Used anti-inflammatory drugs for more than 7 days cumulatively in the last 2 months, or used immunosuppressive drugs, such as corticosteroids; (7) Suffering from chronic infectious or autoimmune diseases, such as lupus, enteritis, hepatitis, etc.; (8) A history of substance dependence or substance abuse.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — identify according to the biological sex
Enrollment: 52 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the change in scores of HAMD-17 after treatment | 4 weeks (at the end week 4)

SECONDARY OUTCOMES:
the change in scores of HAMD-17 after follow up | 12 weeks (at the end week 12)
the change in levels of serum biomarkers after treatment and follow up | 4 and 12 weeks (at the end week 4 and 12)
the change in power of EEG activity in specific brain regions after treatment and follow up | 4 and 12 weeks (at the end week 4 and 12)

CONTACTS AND LOCATIONS:
Locations (1):
- The 20th ward of general psychiatric department, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared if the participants agree.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 2 years after the whole study finished